CLINICAL TRIAL: NCT03959787
Title: Improving Surgical Patient Knowledge and Safe Use of Opioids - a Randomized Controlled Trial
Brief Title: Surgical Patient Knowledge and Safe Use of Opioids
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Ontario Ministry of Health and Long Term Care (Other Government)
Responsible Party: Principal Investigator, Jean Wong, Principal Investigator, University Health Network, Toronto
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Version 15-April-2019
Record Dates: First submitted 2019-05-11; First posted 2019-05-22 (Actual); Last update posted 2021-10-28 (Actual); Status verified 2021-10

CONDITIONS: Opioid Use

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Educational pamphlet and standard care (Experimental): patients randomized to the educational pamphlet arm will receive the educational pamphlet
  Interventions: Other: Educational
- control group - standard care (No Intervention): Patients randomized to control arm, will receive the standard care.

INTERVENTIONS:
Other: Educational — Educational pamphlet will be given to intervention group.
  Arms: Educational pamphlet and standard care

SUMMARY:
Opioids are commonly prescribed for surgical patients to treat moderate to severe pain after surgery. However, opioids can be associated with serious complications such as respiratory depression and death. Currently, it is not routine practice to provide standardized written materials to surgical patients about the risks of opioids and how to safely use opioids after surgery. Investigator has developed an educational pamphlet specifically for surgical patients to educate them about the safe use of opioids.

The objective of this study is to determine whether the pamphlet increases surgical patients' knowledge about the safe use, proper storage and disposal of opioids.

DETAILED DESCRIPTION:
Participants presenting to the preoperative clinic will be recruited for this trial. After informed consent is obtained, patients will be randomized to one of 2 groups: 1) educational pamphlet and standard care, or 2) control group - standard care (no pamphlet) All patients will complete the opioid knowledge questionnaire to test baseline knowledge on opioids. If patient is randomized to the educational pamphlet and standard care, patient will receive the educational pamphlet and standard care. After the patient reviews the pamphlet, the patient will complete the questionnaire again. If the patient is randomized to the control group, the patient will receive the usual standard of care.

All patients will be contacted by telephone 15 days and 30 days after surgery to conduct the follow-up.

ELIGIBILITY:
Inclusion Criteria:

* All English speaking
* Adult (≥18 yrs) surgical patients presenting to the Preoperative Clinic

Exclusion Criteria:

* Patients who are on opioids for chronic pain
* Patients have taken opioids in the past 30 days
* Patients who are unable to read and understand English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2019-05-23 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Change in knowledge | day 1
  Change in knowledge on safe opioid use questionnaire immediately post-education.

SECONDARY OUTCOMES:
Knowledge retention | 15 and 30 days
  Knowledge retention of safe opioid use questionnaire 15 days/30 days post-education. Proper disposal of unused opioids.

CONTACTS AND LOCATIONS:
Overall Officials: Jean Wong, MD, Principal Investigator — University Health Network, Toronto
Locations (2):
- Canada (2):
  - Women's College Hospital, Toronto, Ontario
  - Toronto Western Hospital, University Health Network, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No